CLINICAL TRIAL: NCT02738255
Title: Effect of Added Varnum Mouthpiece on Pharyngeal Collapsibility and Sleep Apnea Severity in Mouth Breathers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Andrew Wellman (Other)
Responsible Party: Sponsor-Investigator, David Andrew Wellman, Associate Professor, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012P000957F
Record Dates: First submitted 2016-04-12; First posted 2016-04-14 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Mouth breathing; Apnea-Hypopnea Index (AHI)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Mouth Breathing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polysomnogram With Varnum First, Regular Polysomnogram Second (Active Comparator): Varnum mouthpiece, similar to a mouth tape with central opening on the first night, then a 1-week non-treatment period, then overnight sleep study with no mouthpiece.
  Interventions: Device: Varnum mouthpiece
- Regular Polysomnogram First, Polysomnogram With Varnum Second (Active Comparator): Baseline sleep study without Varnum mouthpiece on the first night, then a 1-week non-treatment period, then an overnight sleep study with Varnum mouthpiece on the second night.
  Interventions: Device: Varnum mouthpiece

INTERVENTIONS:
Device: Varnum mouthpiece — An adhesive mouthpiece with a central opening applied during sleep
  Other Names: Somnifix mouthpiece

SUMMARY:
Test the effect of added a single-use Varnum mouthpiece on pharyngeal collapsibility and obstructive sleep apnea (OSA) severity in patients who identify themselves as mouth breathers. Research indicates that nasal breathing not only may improve sleep apnea but it also increases circulation, blood oxygen, and carbon dioxide levels, slows the breathing rate, and improves overall lung volumes. Thus, the investigators will test whether a single-use Varnum mouthpiece can improve pharyngeal collapsibility and OSA severity in mouth breathers.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder that remains under-treated due few therapeutic options beyond continuous positive airway pressure (CPAP). In patients with OSA, upper airway obstruction is caused by collapse of pharyngeal structures during sleep. It is known that mouth breathing increases upper-airway collapsibility during sleep and may contribute to the occurrence of sleep disordered breathing. In addition, it was shown that patients with a high percentage of mouth breathing during sleep were less adherent to CPAP therapy. Therefore, one potential solution to these problems is to use Varnum's mouthpiece to prevent mouth breathing during sleep.

The overall objective of the current study is to improve upper airway collapsibility and sleep apnea in OSA patients who have a high percentage of mouth breathing during sleep. The investigators' central hypothesis is that preventing the lips from parting with the Varnum device will reduce oral breathing and thereby OSA severity in mouth breathers. The investigators chose this hypothesis because "taping the mouth closed" with a simple device such as the Varnum mouthpiece is the most straightforward approach to dealing with this common problem. With this research, it could become possible to overcome one of the major problems contributing to sleep apnea - mouth breathing.

Therefore, the investigators aim to test the effect of the Varnum mouthpiece on pharyngeal collapsibility and OSA severity in patients who identify themselves as mouth breathers. The investigators' working hypothesis is that the device will keep the lips from separating and thereby prevent oral breathing. In doing so, it may help keep the airway more patent (by promoting nasal instead of oral breathing) in self-described mouth breathers and thus reduce OSA severity. On the contrary, the investigators believe patients who do not identify themselves as mouth breathers might not benefit significantly from the Varnum device.

The expected outcome of this study is validation of new device for improving sleep apnea in a large subgroup of easily identifiable OSA patients, namely self-described mouth breathers. Such a device could advance the field by providing more effective alternative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Presence of obstructive sleep apnea (AHI>10 events/hr)

Exclusion Criteria:

* Serious co-morbidities including lung disease, heart disease, renal disease
* Medications affecting respiration or sleep

Mouth breather subgroup inclusion criteria: self-described mouth breathing habit during sleep.

non-mouth breathing subgroup inclusion criteria: absence of self-described mouth breathing during sleep

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polysomnogram With Varnum First, Regular Polysomnogram Second | Regular Polysomnogram First, Polysomnogram With Varnum Second
Started | 11 | 15
Completed | 11 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polysomnogram With Varnum First, Regular Polysomnogram Second | Regular Polysomnogram First, Polysomnogram With Varnum Second | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (13.4) | 55.3 (8.1) | 54.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 7 | 11 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 15 | 26
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: Events/hour] — Apnea-Hypopnea Index (AHI) is the metric used to diagnose and quantify the severity of sleep apnea. AHI measures the frequency of partial and complete airway obstructions during sleep.
  Events/hour | 17.0 (14.3) | 25.5 (18.1) | 21.9 (16.8)
Snoring Index [Mean (Standard Deviation); unit: Events/hour] — Snoring Index quantifies the number of breaths with snoring per hour of sleep. This was only measured in simple snorers who had an apnea-hypopnea index <10 events/hour Population: Only simple snorers with AHI<10 were analyzed for this outcome
  Events/hour
    number analyzed (Participants) | 5 | 3 | 8
    (all) | 36.0 (57.9) | 331.2 (271.7) | 146.7 (215.3)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Apnea Severity as Measured by Apnea-hypopnea Index (AHI)
Description: The number of respiratory events (apneas and hypopneas) per hour of sleep. This was measured on two nights in random order (night with Varnum mouthpiece and night without Varnum mouthpiece). The median AHI on the night with Varnum mouthpiece was then compared with median AHI on the night without Varnum mouthpiece.
Time Frame: Two nights: night with Varnum mouthpiece and night without Varnum mouthpiece
Measure: Median (Inter-Quartile Range); unit: Events/hour
Groups:
- Polysomnogram With Varnum Mouthpiece: Varnum mouthpiece, similar to a mouth tape with central opening
- Regular Polysomnogram: Overnight sleep study without Varnum mouthpiece
Arm/Group | Polysomnogram With Varnum Mouthpiece | Regular Polysomnogram
Number analyzed (Participants) | 25 | 25
Events/hour | 16.4 [2.1 to 34.7] | 15.8 [1.1 to 29.9]

2. Secondary Outcome: Pharyngeal Collapsibility as Measured by Median Peak Inspiratory Flow During Sleep
Description: The median peak flow during sleep was measured and compared on both nights (night with Varnum mouthpiece and night without Varnum mouthpiece). The median peak flow is a surrogate measure of upper airway collapsibility.
Time Frame: Two nights: night with Varnum mouthpiece and night without Varnum mouthpiece
Measure: Median (Inter-Quartile Range); unit: L/s
Groups:
- Polysomnogram With Varnum Mouthpiece: Median peak flow from the night with Varnum mouthpiece
- Regular Polysomnogram: Median peak flow from the night without Varnum mouthpiece
Arm/Group | Polysomnogram With Varnum Mouthpiece | Regular Polysomnogram
Number analyzed (Participants) | 25 | 25
L/s | 0.32 [0.10 to 0.40] | 0.36 [0.16 to 0.39]

3. Secondary Outcome: Snoring Index in Simple Snorers
Description: Snoring index is the number of breaths with snoring per hour of sleep. This was measured in both nights (night with Varnum mouthpiece and night without Varnum mouthpiece) only in simple snorers with AHI<10. The median of snoring index was compared between night with Varnum mouthpiece and night without Varnum mouthpiece.
Time Frame: Two nights: night with Varnum mouthpiece and night without Varnum mouthpiece
Population: This outcome was only calculated for simple snorers with AHI<10 events/hour.
Measure: Median (Inter-Quartile Range); unit: Snore/hour
Groups:
- Polysomnogram With Varnum Mouthpiece: Number of snores per hour on the night with Varnum mouthpiece
- Regular Polysomnogram: Number of snores per hour on the night without Varnum
Arm/Group | Polysomnogram With Varnum Mouthpiece | Regular Polysomnogram
Number analyzed (Participants) | 8 | 8
Snore/hour | 3.0 [1.0 to 10.6] | 30.4 [12.3 to 198.8]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Three types of adverse event data are reported, including "All-Cause Mortality," "Serious," and "Other (Not Including Serious)" Adverse Events.
Arm/Group | Polysomnogram With Varnum Mouthpiece | Regular Polysomnogram
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02738255/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02738255/SAP_001.pdf